CLINICAL TRIAL: NCT05513443
Title: Prostate Cancer IRE Study (PRIS) - A Randomized Controlled Trial Comparing Focal to Radical Treatment in Localized Prostate Cancer
Brief Title: Prostate Cancer IRE Study (PRIS)
Acronym: PRIS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Anna Lantz, MD PhD Principal Investigator Associate Professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: K2021-4853; 4-1421/2022 (Other: Karolinska Institutet)
Record Dates: First submitted 2022-08-17; First posted 2022-08-24 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2025-01

CONDITIONS: Prostate Cancer
Keywords: Focal treatment; IRE
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Electroporation; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- PRIS 1, arm 1 (Experimental): Men randomized to the experimental arms will be offered focal treatment of prostate cancer with IRE technology. IRE stands for "irreversible electroporation" and involves the use of high voltage electrical pulses to treat solid tumors by increasing membrane permeability and inducing membrane disruption, leading to cell death.
  Interventions: Procedure: Irreversible electroporation, IRE
- PRIS 1, arm 2 (Active Comparator): Men eligible for radical prostatectomy and randomized to the control arm will undergo radical prostatectomy in line with national guidelines.
  Interventions: Procedure: Radical prostatectomy
- PRIS 2, arm 1 (Experimental): Men randomized to the experimental arms will be offered focal treatment of prostate cancer with IRE technology. IRE stands for "irreversible electroporation" and involves the use of high voltage electrical pulses to treat solid tumors by increasing membrane permeability and inducing membrane disruption, leading to cell death.
  Interventions: Procedure: Irreversible electroporation, IRE
- PRIS 2, arm 2 (Active Comparator): Men eligible for radiation therapy and randomized to the control arm will undergo radiation therapy in line with national guidelines.
  Interventions: Radiation: Radiation therapy

INTERVENTIONS:
Procedure: Irreversible electroporation, IRE — IRE involves the use of high voltage electrical pulses to treat solid tumors by increasing membrane permeability and inducing membrane disruption, leading to cell death. The technique is used in Sweden today in radical ablative therapies in the treatment of tumors in the liver, kidney and pancreas. Prior to treatment a Foley catheter is placed. During the treatment, which takes place under anesthesia, the patient is placed in gynecological position and the tumour lesion is located with BK transrectal fusion ultrasound. Thereafter the needles are placed transperineal around the tumor in the prostate using a brachytherapy grid (17Ga Civco brachytherapy grid), guided by the ultrasound/MRI fusion images. Through the needles electrical pulses are then sent to treat the tumor in the center using the Nanoknife technique. After treatment patients are treated with diuretics to flush the kidneys post treatment.
  Arms: PRIS 1, arm 1; PRIS 2, arm 1
Procedure: Radical prostatectomy — Radical prostatectomy
  Arms: PRIS 1, arm 2
Radiation: Radiation therapy — Radiation therapy for prostate cancer
  Arms: PRIS 2, arm 2

SUMMARY:
The aim of this study is to evaluate the feasibility to treat localized prostate cancer diagnosed with MRI and targeted/systematic biopsies, with IRE in comparison with conventional radical treatments with the primary objective to locally control the tumour with a minimum of side effects.

DETAILED DESCRIPTION:
OBJECTIVES The aim of the proposed research is to evaluate the cancer control, genitourinary, rectal and overall health-related quality of life outcomes of focal therapy for unifocal localized prostate cancer using irreversible electroporation (IRE).

PRIMARY AIM

• To evaluate functional outcomes in men treated for unifocal ISUP 2-3 localized prostate cancer with focal treatment in comparison to conventional treatment with either radical prostatectomy or radiation therapy

SECONDARY AIMS

* To evaluate adverse events in men treated for unilfocal ISUP 2-3 localized prostate cancer with focal treatment in comparison to conventional treatment with either radical prostatectomy or radiation therapy
* To evaluate progression free and treatment free survival in men treated for unifocal ISUP 2-3 localized prostate cancer with focal treatment in comparison to conventional treatment with either radical prostatectomy or radiation therapy
* Economic evaluation of each technique

TRIAL DESIGN This study is a randomized controlled exploratory trial comparing focal therapy to conventional radical treatment of prostate cancer with the primary aim to evaluate functional outcomes 12 months after treatment.

Patients will be included from 4 different hospitals within the Stockholm County; Karolinska University Hospital, Danderyd Hospital, St Görans Hospital, Södersjukhuset. Eligible patients, after MRI and targeted/systematic biopsies, will be men with clinically significant intermediate-risk PCa or dominant unifocal clinically significant intermediate-risk and small contralateral low-risk disease without previous history of prostate cancer treatment.

Potential study participants will have a visit scheduled together with an urologist and oncologist, where a treatment decision of radical prostatectomy or radiation therapy will be done together with the patient. At this visit the patient will receive oral and written information about the study. If the patient is interested in participating, a baseline visit is scheduled during which informed consent is obtained and the patient randomized to one of two standard treatments or focal treatment.

Patients eligible for radical prostatectomy will be randomized in study 1 to focal treatment or radical prostatectomy. Patients eligible for radiation therapy will be randomized in study 2 to focal treatment or radiation therapy. Time between randomization and treatment will be <= 6 weeks.

Patients will be asked to fill out study specific questionnaires with questions on functional outcomes and quality of life.

Main outcome measurement in study 1 will be urinary incontinence at 12 months post treatment and in study 2 irritative urinary symptoms 12 months post treatment. Further outcomes will be erectile dysfunction, adverse events, progression-free and treatment-free survival.

ELIGIBILITY:
Inclusion Criteria:

* Age at inclusion ≥ 40 years
* MRI-visible lesion

  * EPE 3* <1.5 cubic cm3 lesion volume
* Gleason score 3 + 4 or 4 + 3 from a single MRI-visible lesion without any Gleason grade 4 in systematic biopsies outside of the target
* PSA level ≤ 20 ng/ml
* Clinical stage ≤ T2c disease
* Unifocal significant disease
* Life expectancy of ≥ 10 years
* Sufficient proficiency in the Swedish language to understand written and verbal information about the trial, its consent process and the study questionnaires

  * Extraprostatic extension; 5-grade Likert scale 1=

Exclusion Criteria:

* Intraductal tumour
* History of treatment for prostate cancer; surgery, radiation, chemotherapy or hormonal treatment
* History of cardiac arrythmias
* Pacemaker
* Renal insufficiency; GFR<30
* Severe illnesses such as concomitant cancers, severe cardio-vascular disease or dementia
* Contraindications for magnetic resonance imaging (MRI) e.g. magnetic cerebral clips, cochlear implants or severe claustrophobia
* History of bladder cancer
* History of previous pelvic radiotherapy

Min Age: 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Primary outcome in PRIS 1: Urinary continence | 12 months postoperatively
  Urinary incontinence defined by Q3 in EPIC-26, ≥1 pad/day ("Yes") versus none ("No")
Primary outcome in PRIS 2: Irritative urinary symptoms | 12 months postoperatively
  Irritative urinary symptoms defined by Q4e in EPIC-26, Moderate/big problem ("Yes") Versus no/small problem ("No")

SECONDARY OUTCOMES:
Erectile dyfunction | 12 months postoperatively
  IIEF score: International Index of Erectile Function, change. The possible scores for the IIEF-5 range from 5 to 25, and ED was classified into five categories based on the scores: severe (5-7), moderate (8-11), mild to moderate (12-16), mild (17-21), and no ED (22-25).
Voiding function | 12 months postoperatively
  International Prostate Symptom Score (IPSS score), change. It is a validated, reproducible scoring system to assess disease severity and response to therapy. The IPSS is made up of 7 questions related to voiding symptoms. A score of 0 to 7 indicates mild symptoms, 8 to 19 indicates moderate symptoms and 20 to 35 indicates severe symptoms.
Bowel function | 12 months postoperatively
  Expanded Prostate Cancer Index, EPIC-26, Q6 change in score. The EPIC-26 is a validated instrument that measures health-related quality of life across 5 PCa-specific domains. Consequently, the minimum symptom score (best HRQOL) = 0 and the maximum symptom score (worst HRQOL) = 12 in each domain. For consistency, the values assigned to each question range from 0 (best) to 4 (worst) regardless of whether there were 4 or 5 response options per question.
Adverse events | 3 months postoperatively
  Clavien-Dindo
Quality of life, EuroQoL-5 Dimensions | 12 months postoperatively
  EQ5D; The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems.
Treatment Failure, experimental arms | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months
  1. Need for additional focal or whole gland treatment or ADT
  2. Need for whole gland treatment or ADT
  3. Need for whole gland treatment or ADT or ISUP 2 at 12 mo biopsy
Treatment Failure, control arm (surgery) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months
  Post-operative PSA ≥0.2 ng/ml or adjuvant treatments including ADT
Treatment Failure, control arm (radiation) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months
  PSA >2 over nadir (Phoenix) or adjuvant treatments including ADT

CONTACTS AND LOCATIONS:
Overall Officials: Anna Lantz, Ass Prof, Principal Investigator — Karolinska University Hospital and Karolinska Institutet
Locations (1):
- Karolinska Institutet, Stockholm, Solna, Sweden

IPD SHARING:
Plan to Share IPD: No